CLINICAL TRIAL: NCT07258082
Title: Transauricular Vagus Nerve Stimulation (taVNS) for Delirium
Brief Title: TaVNS for Delirium
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Isadora Botwinick, Clinical Assistant Professor of Surgery, Stony Brook University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: IRB2025-00131
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Delirium Treatment; Delirium
Keywords: delirium; tavns; transauricular vagus nerve stimulation; vagus nerve stimulation; transcutaneous vagus nerve stimulation
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- TaVNS and Usual Care for Delirium (Experimental): Hospitalized, right-hand-dominant adults (age ≥ 22) with delirium, receive transauricular vagus nerve stimulation (taVNS) in addition to standard clinical management. TaVNS is administered twice a day, for a maximum of 7 days, until delirium resolves or the patient is discharged from the ICU.
  Interventions: Device: Transauricular Vagus Nerve Stimulation

INTERVENTIONS:
Device: Transauricular Vagus Nerve Stimulation — TaVNS starts within 24 hours of consent and is given twice daily (~30 minutes per session, ≥6 hours apart) for up to 7 days or until delirium resolves. Stimulation will be delivered to the tragus of the left ear via non-invasive clip-on electrode.
  Stimulation parameters will be set to: pulse width 500 µs, frequency 25 Hz, 30 s on / 30 s off. Current amplitude will be titrated to perceptual threshold (0.5-5.0 mA); if patients are unable to participate in perceptual threshold titration, then 1.25 mA will be utilized. On the first day of stimulation, patients will undergo 10 minutes of baseline EEG and cerebral oximetry, followed by 10 minutes of EEG and cerebral oximetry during taVNS.

SUMMARY:
The goal of this clinical trial is to test whether a non-invasive device called transauricular vagus nerve stimulation (taVNS) is safe, practical, and potentially helpful for patients in the hospital who develop delirium. Delirium is a state of confusion that often happens to people in the hospital who are sick or hurt. It can cause agitation, trouble paying attention and difficulty understanding what is happening. Delirium may slow overall recovery.

This study will focus on feasibility and safety. Researchers want to learn whether taVNS can be given safely to critically-ill patients, whether patients and staff can tolerate the treatments, and whether the device produces measurable changes in brain activity and brain oxygen levels.

The main questions this study aims to answer are:

* Is it possible to deliver taVNS safely and consistently to patients in the ICU who have delirium?
* Do patients tolerate the device without significant side effects or complications?
* Does taVNS cause short-term changes in brain signals and oxygen levels that may suggest effects on brain function? This is an early feasibility study and there is no randomization or placebo group. All patients enrolled will receive taVNS in addition to their usual hospital care for delirium.

What participants will do:

* Be identified by their hospital care team and have a confirmed diagnosis of delirium.
* Provide consent (or have a legally authorized representative provide consent if the patient cannot.)
* Undergo brief assessments of thinking and attention (for example, the CAM-ICU test.)
* Receive taVNS treatment using a small clip electrode placed on the ear.

  * The device sends gentle electrical pulses to the nerve in the ear.
  * Each session lasts about 30 minutes, given twice per day (morning and evening, with at least 6 hours between sessions).
  * Treatment can continue for up to 7 days while the patient is in the ICU.
* Be monitored during and after each session. The study team will check vital signs, examine the ear for irritation, and ask about any discomfort.
* On the first day, researchers will also record brain signals (EEG) and brain oxygen levels before and during stimulation using FDA-approved hospital monitoring devices.

Possible risks and discomforts:

* Mild side effects are possible, such as tingling, a tickling or pricking feeling in the ear, or temporary skin redness where the clip is placed.
* Serious side effects are not expected, but all patients will be closely monitored during and after each session to ensure safety.

Possible benefits:

• Patients may or may not experience personal benefit. The main benefit is helping researchers learn whether this treatment approach is safe and practical. In the future, taVNS could potentially become a new tool to help treat or prevent delirium in hospitalized patients.

Study size and duration:

* The study will enroll a limited number of ICU patients with delirium at Stony Brook University Hospital.
* Patients may take part for up to 7 days while hospitalized.

Who can join:

* Right-handed, adult patients in the ICU who are diagnosed with delirium.
* People with certain medical conditions (such as brain bleeds, new strokes, pacemakers or other contraindications) may not be able to participate, for safety reasons.

DETAILED DESCRIPTION:
This will be a single-arm, open-label trial to assess the brain blood oxygen saturation and EEG of hospitalized patients with delirium, and to assess feasibility and safety of transauricular vagus nerve stimulation (taVNS) in this population. This is an early feasibility study and there is no randomization or placebo group. All patients enrolled will receive taVNS in addition to usual hospital care for delirium. We aim to recruit 10 patients. Patients will be recruited from an inpatient population in the ICU or hospital unit. Candidates will be identified on daily rounds by a primary medical team. A diagnosis of delirium will be confirmed by a physician trained in psychiatry, neurology or neurocritical care. After inclusion and exclusion are reviewed, a baseline assessment of delirium through the CAM-ICU (Confusion Assessment Method for Intensive Care Unit) will be completed. After screening and informed consent, the patient will be considered as entered into the study. The patient will begin taVNS within 24 hours of enrollment. Patients who are consented but do not begin taVNS within 24 hours will require repeat screening to evaluate updates to clinical condition and repeat CAM-ICU score to ensure they continue to meet inclusion criteria.

We anticipate that in most situations, a legally authorized representative for the patient will be the initial contact for the study as well as the individual providing consent to the study. If a patient were to meet exclusion criteria after enrollment, they would be ineligible for further participation. Previously collected data prior to the event would still be used for analysis.

The study device is the Soterix Medical Transcutaneous auricular Vagus Nerve Stimulator, for which we have submitted an IDE to the FDA and received nonsignificant risk designation (NSR). The device will be configured with the Soterix Medical RELIfit-Tragus accessory to hook around the ear to deliver stimulation to the auricular branch of the vagus nerve in the tragus of the left ear. TaVNS will be performed on the left side to minimize the already negligible risk of cardiac side effects. The device will be set to a frequency of 25 Hz and pulse width of 500 μs based on previous literature. The intensity will be titrated in the first session to a barely perceptible threshold. Patients unable to cooperate with the titration procedure will have their stimulation intensity set at 1.25 mA.

Vitals, relevant medical history, labs and medication data will be collected from the medical record. Prior to initiation of taVNS on the first day, subjects will undergo 10 minutes of neurophysiological monitoring to determine baseline recording. Cerebral oxygenation, hemodynamics, and EEG will be documented using the Masimo O3/Sedline brain monitoring system, a noninvasive, commercially available brain monitor. The Masimo O3/Sedline device will continue to be used to monitor the patient while undergoing taVNS to record further data for another 10 minutes during the first stimulation session.

Subjects will be prescribed two 30-minute sessions of taVNS stimulation each day with a minimum of 6 hours between sessions for a maximum of 7 days until either delirium resolves, or the patient is discharged.

Upon discontinuation of the study, we will screen the subject for any sensory changes, discomfort, or adverse events, as well as perform an additional CAM-ICU screen. The subject will be discharged without follow-up due to the minimal risk in the study. Risks and adverse events associated with use of the Soterix Medical Transcutaneous auricular Vagus Nerve Stimulator are small. We ensure patients use the device only under supervision by the research team, with proper application, and perform regular skin inspections after each stimulation session. Subjects will be supervised during monitoring by study personnel who will observe for any evidence of subject discomfort from monitoring. A member of the study team who is a Stony Brook University Hospital ICU attending intensivist will be present throughout each stimulation session, as well as for the initial device intensity titration. A review of pre- and post-session relevant clinical data (including vitals, medications, skin inspection and labs) will be performed.

All enrolled patients who receive at least one session of taVNS will be included in the final analysis. Patients with incomplete data will be reported and analyzed using available data only, without imputation. Due to the nature of ICU care, compliance with the protocol will be defined as completing at least 1 stimulation session during the 7-day study period.

ELIGIBILITY:
Inclusion Criteria:

* Stony Brook University Hospital inpatient, Age > 22
* Right- handed
* Screen positive for delirium on CAM-ICU instrument

Exclusion Criteria:

* Severe neurologic disability including severe traumatic brain injury, severe permanent cognitive impairment
* Pacemaker present
* Implanted VNS stimulator present
* Personal history of epilepsy
* Facial or ear pain or trauma
* Recent history of substance abuse
* Any other medical condition that, in the judgment of the investigator, makes participation in the study unsafe.
* Weight < 40kg
* Pregnant females
* Intubated patient

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09-26 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility of taVNS in hospitalized patients with delirium | From enrollment to end of treatment at a maximum of 7 days
  We will assess feasibility of taVNS as follows:
  The proportion of stimulation delivered relative to the stimulation prescribed, calculated as:
  Stimulation delivered (minutes) /Stimulation prescribed (minutes)
  Feasibility will be demonstrated if:
  1. The mean proportion of stimulation delivered across the cohort is ≥10%. Previous taVNS studies in adults have demonstrated that as little as 6 minutes of stimulation is adequate to demonstrate neuromodulatory effect as detected by fMRI.
     In our protocol, patients will be prescribed a total of 60 minutes of stimulation per day of study 6 minutes of stimulation (a known minimum effective dose) is thus 10% of prescribed stimulation time.
  2. At least 80% of patients achieve ≥10% of prescribed stimulation.
Feasibility of taVNS in delirious hospitalized patients | From enrollment to the end of study at a maximum of 7 days
  We will assess feasibility of taVNS as follows:
  The proportion of stimulation delivered relative to the stimulation prescribed, calculated as: Stimulation delivered (minutes) / Stimulation prescribed (minutes)
  Feasibility will be demonstrated if:
  1. The mean proportion of stimulation delivered across the cohort is ≥10%. Previous taVNS studies in adults have demonstrated that as little as 6 minutes of stimulation is adequate to demonstrate neuromodulatory effect as detected by fMRI.
     In our protocol, patients will be prescribed a total of 60 minutes of stimulation per day of study. 6 minutes of stimulation (a known minimum effective dose) is thus 10% of prescribed stimulation time.
  2. At least 80% of patients achieve ≥10% of prescribed stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Isadora Botwinick, MD, Principal Investigator — Stony Brook University Hospital
Locations (1):
- Stony Brook University Hospital, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD and supporting information will be available starting 6 months after publication.

REFERENCES:
- [Background] Wilson JE, Mart MF, Cunningham C, Shehabi Y, Girard TD, MacLullich AMJ, Slooter AJC, Ely EW. Delirium. Nat Rev Dis Primers. 2020 Nov 12;6(1):90. doi: 10.1038/s41572-020-00223-4. PMID 33184265
- [Background] Huffman WJ, Subramaniyan S, Rodriguiz RM, Wetsel WC, Grill WM, Terrando N. Modulation of neuroinflammation and memory dysfunction using percutaneous vagus nerve stimulation in mice. Brain Stimul. 2019 Jan-Feb;12(1):19-29. doi: 10.1016/j.brs.2018.10.005. Epub 2018 Oct 9. PMID 30337243
- [Background] Badran BW, Dowdle LT, Mithoefer OJ, LaBate NT, Coatsworth J, Brown JC, DeVries WH, Austelle CW, McTeague LM, George MS. Neurophysiologic effects of transcutaneous auricular vagus nerve stimulation (taVNS) via electrical stimulation of the tragus: A concurrent taVNS/fMRI study and review. Brain Stimul. 2018 May-Jun;11(3):492-500. doi: 10.1016/j.brs.2017.12.009. Epub 2017 Dec 29. PMID 29361441
- [Background] Hshieh TT, Fong TG, Marcantonio ER, Inouye SK. Cholinergic deficiency hypothesis in delirium: a synthesis of current evidence. J Gerontol A Biol Sci Med Sci. 2008 Jul;63(7):764-72. doi: 10.1093/gerona/63.7.764. PMID 18693233